CLINICAL TRIAL: NCT03896165
Title: Teaching Parents Reiki for Their Adolescents Receiving Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Akron Children's Hospital (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018X0079; U2CNR014637 (NIH)
Record Dates: First submitted 2019-03-25; First posted 2019-03-29 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Palliative Care; Chronic Disease
Keywords: Complementary Health Approach; Parent; Adolescent
MeSH Terms: conditions — Chronic Disease | interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Mixed methods quasi-experimental one group design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teaching Reiki (Experimental): Parent-adolescent pairs will be in the study for a total of nine weeks from enrollment to the follow up visit. During Week 1, the parent will receive Reiki training, a poster with suggested hand positions and a commercially-available book about Reiki in the home. During Week 2 the parent will receive a Reiki booster session with a repeat of the training and may ask questions in the home. At the end of Week 4, measures will be repeated either in person or by phone. During Week 8, measures will be repeated, another hair sample obtained and the parent will participate in a qualitative interview. The qualitative interview will be administered in person by trained Ohio State University College of Nursing study staff as part of the interview session. Interviews will be audio recorded using a hand-held audio recording device. Audio recording is voluntary and participants can choose to not have their interview recorded and still be a part of the study.
  Interventions: Other: Reiki

INTERVENTIONS:
Other: Reiki — Reiki is a complementary health approach where trained providers place their hands lightly on or just above a person, in discrete positions, with the goal of facilitating the person's own healing response. A Reiki practitioner will perform the initial teaching and instruct the parent how to perform a simple 15-minute Reiki session. Parents will complete a return demonstration using light touch with their adolescent. Parents will be asked to complete a minimum of 15 minutes of Reiki with their adolescent at least five days per week for the four-week intervention period.

SUMMARY:
The proposed study addresses National Institute of Nursing Research (NINR) priorities of advancing symptom science to "develop [and] test … novel, scalable symptom management interventions, including complementary health approaches (CHAs), in real-world clinical settings to improve health outcomes and quality of life" and the science of compassion to improve palliative and end-of-life care through "developing, testing, and implementing personalized, culturally congruent, and evidence-based palliative and hospice interventions that best address the needs of underserved, disadvantaged, and diverse populations across the care continuum." A long-term bonus of teaching parents to deliver Reiki is that Reiki is highly scalable and once learned, costs nothing to use, an important potential overall cost savings over other CHAs.

DETAILED DESCRIPTION:
Despite advances in the assessment and treatment of symptoms, including pain in adolescents receiving palliative care, parents still report that their children suffer. Advances in medical science and care have led to a growing number of children living with life-limiting chronic conditions. Out of 83 million children under the age of 19,16 an estimated 600,000 to 1,600,00017 are living with life-threatening/life-limiting conditions and over 180,000 are considered "medically fragile." These children require intense medical and nursing care in the home and often experience lengthy, recurrent hospital stays, accounting for about 26% of hospital days and 41% of hospital charges. Adolescents with life-threatening/life-limiting conditions, many of whom are developmentally delayed, experience many symptoms and have complex co-morbidities requiring medical management.

Many of these adolescents could benefit from complementary health approaches (CHAs) such as Reiki, a gentle light touch biofield energy therapy. Parents of adolescents receiving palliative care also experience high levels of stress. Previous studies have shown that empowering parents in the care of their chronically ill child help parents better cope with challenges. Some CHAs show promise for symptom management without side effects, such as sedation from additional medication, thereby permitting greater alertness and allowing more interaction with family and friends. Preliminary evidence from the PIs pilot study showed that professionally-delivered Reiki is feasible for children and adolescents receiving palliative care at home. The majority of parents said they wished they could learn Reiki so they might provide this relaxing therapy in the moment it was needed rather than waiting for the next professional session. One non-experimental program found that teaching parents Reiki was feasible and acceptable in the hospital. Parents who participated in two or more training sessions felt more confident providing Reiki. During informal interviews, parents said they felt good at being an active participant in their child's care and that their child experienced increased comfort, relaxation, and decreased pain.

Parents of disabled adolescents receiving palliative care often suffer from high caregiver burden and chronic stress leading to co-morbidities and decreased QoL. A cross-sectional survey conducted in Europe examined stress in 818 parents caring for a child with cerebral palsy. Results showed that 26% of mothers had very high stress. When the child had a communication or intellectual impairment or moderate-to-severe pain, parental stress was higher. One study examined psychological burden for 204 parents of children with serious chronic conditions. This study found that 75% of parents reported depression, and 67% had anxiety. The investigators are interested in exploring whether adding a skill (Reiki) aimed at decreasing symptoms in the adolescent will result in a decrease in symptoms and chronic stress for the parent.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include adolescent-parent dyads. Dyads will be included if the
* Adolescent: (1) is 10 to 19 years old, (2) is receiving palliative care at home, (3) understands English
* Parent: (1) provides care for the adolescent most days of the week and (2) is able to read and write English at the 6th grade level.

Exclusion Criteria:

* if (1) either the adolescent or the parent are taking or have taken corticosteroids within the last 30 days (affects the hair cortisol levels), or (2) either the adolescent or the parent has less than one inch of hair.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Thrane, PhD, RN, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Akron Children's Hospital, Akron, Ohio
  - The Ohio State University College of Nursing, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Teaching Reiki: Parent-adolescent pairs will be in the study for a total of nine weeks from enrollment to the follow up visit. During Week 1, the parent will receive Reiki training, a poster with suggested hand positions and a commercially-available book about Reiki in the home. During Week 2 the parent will receive a Reiki booster session with a repeat of the training and may ask questions in the home. At the end of Week 4, measures will be repeated either in person or by phone. During Week 8, measures will be repeated, another hair sample obtained and the parent will participate in a qualitative interview. The qualitative interview will be administered in person by trained Ohio State University College of Nursing study staff as part of the interview session. Interviews will be audio recorded using a hand-held audio recording device. Audio recording is voluntary and participants can choose to not have their interview recorded.
  Reiki: Reiki is a complementary health approach where trained providers place their hands lightly on or just above a person, in discrete positions, with the goal of facilitating the person's own healing response. A Reiki Master will perform the initial teaching and instruct the parent how to perform a 15-minute Reiki session. Parents will complete a return demonstration using light touch with their adolescent. Parents will be asked to complete a minimum of 15 minutes of Reiki with their adolescent at least five days per week for the four-week intervention period.
Period: Overall Study
Arm/Group | Teaching Reiki
Started | 20
Completed | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Ten parent-adolescent pairs (20 participants total)
Groups:
- Teaching Reiki: Parent-adolescent pairs will be in the study for a total of 9 weeks from enrollment to the follow up. Week 1, the parent will receive Reiki training, a poster with suggested hand positions and a commercially-available book about Reiki in the home. Week 2 the parent will receive a Reiki booster session with a repeat of the training and asking questions in the home. At the end of Week 4, measures will be repeated either in person or by phone. Week 8, measures will be repeated, another hair sample obtained and the parent will participate in a qualitative interview. The qualitative interview will be administered in person by trained Ohio State University College of Nursing study staff. Interviews will be audio recorded using a hand-held audio recording device. Audio recording is voluntary and participants can choose to not have their interview recorded and still be a part of the study.
  Reiki: Reiki is a complementary health approach where trained providers place their hands lightly on or just above a person, in discrete positions, with the goal of facilitating the person's own healing response. A Reiki practitioner will perform the initial teaching and instruct the parent how to perform a simple 15-minute Reiki session. Parents will complete a return demonstration using light touch with their adolescent. Parents will be asked to complete a minimum of 15 minutes of Reiki with their adolescent at least five days per week for the four-week intervention period.
Arm/Group | Teaching Reiki
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 10 parent-adolescent pairs (10 parents and 10 adolescents for a total of 20 participants)
  years
    Adolescent: number analyzed (Participants) | 10
    Adolescent | 14.0 (3.16)
    Parent: number analyzed (Participants) | 10
    Parent | 47.2 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction of Parents Learning Reiki in the Home to Use With Their Adolescent Receiving Palliative Care.
Description: Satisfaction will be examined by computing the proportion of approached subjects who enroll in the study, the proportion of subjects who complete Reiki training, and the proportion of enrolled subjects who complete data collection.
Time Frame: Four weeks
Population: Number of enrolled participants who completed Reiki training activities
Measure: Count of Participants; unit: Participants
Groups:
- Teaching Reiki: Parent-adolescent pairs will be in the study for a total of 9 weeks from enrollment to the follow up visit. Week 1, the parent will receive Reiki training, a poster with suggested hand positions and a commercially-available book about Reiki in the home. Week 2 the parent will receive a Reiki booster session with a repeat of the training and may ask questions in the home. At the end of Week 4, measures will be repeated either in person or by phone. Week 8, measures will be repeated, another hair sample obtained and the parent will participate in a qualitative interview. The qualitative interview will be administered in person by trained Ohio State University College of Nursing study staff. Interviews will be audio recorded using a hand-held audio recording device. Audio recording is voluntary and participants can choose to not have their interview recorded and still be a part of the study.
  Reiki: Reiki is a complementary health approach where trained providers place their hands lightly on or just above a person, in discrete positions, with the goal of facilitating the person's own healing response. A Reiki practitioner will perform the initial teaching and instruct the parent how to perform a simple 15-minute Reiki session. Parents will complete a return demonstration using light touch with their adolescent. Parents will be asked to complete a minimum of 15 minutes of Reiki with their adolescent at least five days per week for the four-week intervention period.
Arm/Group | Teaching Reiki
Number analyzed (Participants) | 20
Participants | 18

2. Secondary Outcome: Rate of Change in Adolescents' and Parents' Stress Response (as Measured by Hair Sample).
Description: Explore the adolescents' and parents' stress response. We will measure hair cortisol at the beginning and again at week 9.
Time Frame: Week 0, week 9
Population: Data was unable to be collected
Arm/Group | Teaching Reiki
Number analyzed (Participants) | 0

3. Secondary Outcome: Rate of Change in Adolescents' and Parents' Stress Response (as Measured by Saliva Alpha Amylase).
Description: We will also measure saliva alpha amylase twice per week for 4 weeks.
Time Frame: Week 1, week 2, week 3, week 4
Population: Data was unable to be collected
Arm/Group | Teaching Reiki
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Adolescents' and Parents' Symptom Profile as Measured by Patient Reported Outcome Measurement Information System (PROMIS) Symptom Questionnaire.
Description: Explore the adolescents' and parents' symptom profile (as measured by changes in physical function, anxiety, depression, fatigue, sleep, social roles, and pain level).
Time Frame: Week 0, Week 4, Week 9
Population: Data was unable to be collected
Arm/Group | Teaching Reiki
Number analyzed (Participants) | 0

5. Secondary Outcome: Explore the Parents Confidence in Delivering Reiki Through Audio-recorded Interviews
Description: Explore parents' confidence in delivering Reiki to their adolescent after completing Reiki training and practicing providing Reiki to their adolescent.
Time Frame: Week 9
Population: Data was unable to be collected
Arm/Group | Teaching Reiki
Number analyzed (Participants) | 0

6. Secondary Outcome: Explore Parents' Confidence Their Ability to Help Their Adolescent Through Audio-recorded Interviews
Description: Explore parents' confidence their ability to help their adolescent after completing Reiki training and practicing providing Reiki to their adolescent.
Time Frame: Week 9
Population: Data was unable to be collected
Arm/Group | Teaching Reiki
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Nine weeks.
Description: All adverse event information collected concurs with the clinicaltrials.gov definitions
Groups:
- Teaching Reiki: Parent-adolescent pairs will be in the study for a total of nine weeks from enrollment to the follow up visit. Week 1, the parent will receive Reiki training, a poster with suggested hand positions and a commercially-available book about Reiki in the home. Week 2 the parent will receive a Reiki booster session with a repeat of the training and may ask questions in the home. At the end of Week 4, measures will be repeated either in person or by phone. Week 8, measures will be repeated, another hair sample obtained and the parent will participate in a qualitative interview. The qualitative interview will be administered in person or over Zoom by trained Ohio State University College of Nursing study staff. Interviews will be audio recorded using a hand-held audio recording device. Audio recording is voluntary and participants can choose to not have their interview recorded and still be a part of the study.
  Reiki: Reiki is a complementary health approach where trained providers place their hands lightly on or just above a person, in discrete positions, with the goal of facilitating the person's own healing response. A Reiki Master will perform the initial teaching and instruct the parent how to perform a 15-minute Reiki session. Parents will complete a return demonstration using light touch with their adolescent. Parents were asked to complete a minimum of 15 minutes of Reiki with their adolescent at least five days per week for the 4-week intervention period.
Arm/Group | Teaching Reiki
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT03896165/Prot_SAP_000.pdf